CLINICAL TRIAL: NCT02445092
Title: Double Blind Randomized Controlled Trial on the Effect of Pre-washing the Insemination Catheter on Pregnancy Outcome
Brief Title: The Effect of Pre-washing the Insemination Catheter on Pregnancy Outcome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After reviewing the interim analysis results the study was terminated as a bigger sample size was needed to find a significant difference between the groups.
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Patricia Monnier, Associate Professor at MUHC reproductive health center, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 13-158-SDR
Record Dates: First submitted 2014-01-08; First posted 2015-05-15 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Infertility; Pregnancy
Keywords: Intrauterine insemination; Insemination catheter prewashing; Pregnancy outcome
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Catheter prewashing (Experimental): Intervention: prewashing the catheter before IUI.
  450 patients randomly included in this group will have their insemination catheter prewashed with the same media used to wash the sperm, prior to performing the insemination using the washed catheter.
  Interventions: Other: washing the insemination catheter with sperm washing media
- Control group (No Intervention): 450 patients randomly assigned in this group will have their insemination performed routinely, without washing the insemination catheter..

INTERVENTIONS:
Other: washing the insemination catheter with sperm washing media — Intervention: pre-washing of the IUI catheter
  Throughout the research period all of the insemination catheters used for patients recruited in our study, will be prepared as follows:
  * Connection: The catheter used for insemination, will be connected to the sperm filled syringe as per our standard procedure.
  * Catheter washing: The sperm washing media will be aspirated and then flushed through the insemination catheter..
  * Sperm loading: catheters washed or not connected to the syringe will be loaded with the washed sperm sample as our standard procedure.
  Labeling:
  Patient identification data will be labeled on the syringe and place back in the original package cover to ensure proper blinding and sterility of the catheter.
  Arms: Catheter prewashing

SUMMARY:
The investigators hypothesize that washing the insemination catheter prior to performing the IUI (intrauterine insemination) will improve the pregnancy outcome in IUI cycles when compared to controls (without pre-washing the catheter).

Catheter washing is performed routinely before embryo transfer, however it is not done for IUI catheters. Therefore no data is available on applying the technique to IUI catheters prior to insemination.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary objective:

To determine if pre-washing the catheter before insemination improves the pregnancy outcome in women undergoing IUI.

Secondary objectives:

1. To evaluate the impact of pre-washing the catheter before insemination on the ectopic pregnancy rate in women undergoing IUI.
2. To evaluate the impact of pre-washing the catheter before insemination on the miscarriage rate in women undergoing IUI.
3. To evaluate the impact of pre-washing the catheter before insemination on the multiple pregnancy rates in women undergoing IUI.

STUDY DESIGN:

The study will be a prospective double blind trial among women undergoing IUI at the MUHC reproductive centre using a cluster randomized design. The week will be defined as the unit for the clusters of randomization. Weeks will be allocated to one of the following groups:

* Group 1 = pre-washing group (patients will have the IUI with a pre-washed catheter during that week)
* Group 2 = control group (no pre-washing before IUI during that week)

A random block size will be used to minimize the risk of non-blinding. The study is double-blind, neither the patients nor the physicians performing IUI will know whether the catheter was washed or not, as both the sample and the catheter will be prepared by the andrology lab technician. The cluster randomization design is justified since the management of the unit will not allow us to perform a randomization at the patient level.

However a very low Intra-Correlation Coefficient (ICC) between patients is expected.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women age ranges from 18 to 40 years at the time of treatment at the MUHC reproductive centre.
* Patients undergoing IUI.
* Fresh and frozen sperm treatment cycles
* Hormone induced and natural cycle (no hormonal stimulation).
* Patients speaking English or/and French.
* Patients able to consent.

Exclusion Criteria:

* Patients younger than 18 years or older than 40 years of age.
* Patients undergoing ovarian stimulation without IUI.
* Patients who have been recruited in our study in a previous IUI cycle.
* Patients who don't speak English or French.
* Patients who are not able or refuse to consent.
* Patient who are recruited in a different IUI research study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2014-01; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Pregnancy Rate | 19months
  To determine if pre-washing the catheter before insemination improves the pregnancy outcome in women undergoing IUI.

SECONDARY OUTCOMES:
Ectopic Pregnancy Rate | 19 months
  1. To evaluate the impact of pre-washing the catheter before insemination on the ectopic pregnancy rate in women undergoing IUI.
Clinical pregnancy rate | 19 months
  2. To evaluate the impact of pre-washing the catheter before insemination on the clinical pregnancy rate in women undergoing IUI.
miscarriage Rate | 19 months
  3. To evaluate the impact of pre-washing the catheter before insemination on the miscarriage rates in women undergoing IUI.
Live birth rate | 19 months
  To evaluate the impact of pre-washing the catheter before insemination on the live birth rates in women undergoing IUI.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Monnier, MD, Principal Investigator — MUHC reproductive center
Locations (1):
- MUHC reproductive center, Montreal, Quebec, Canada

REFERENCES:
- [Background] Pont JC, Patrat C, Fauque P, Camp ML, Gayet V, Wolf JP. [Pre-washing catheter dramatically improves the post intrauterine insemination pregnancy rate]. Gynecol Obstet Fertil. 2012 Jun;40(6):356-9. doi: 10.1016/j.gyobfe.2012.02.002. Epub 2012 Apr 13. French. PMID 22503402